CLINICAL TRIAL: NCT02246036
Title: Clinical Trial to Assess the Tolerance and the Safety of a Duodenal Tube Monitoring the Microcirculation in 10 Critically Ill Patients.
Brief Title: Tolerance and Safety of a Duodenal Probe Monitoring the Microcirculation
Acronym: MC Monitor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Perfusion Diagnostics (Industry)
Collaborators: CEISO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00989-38
Record Dates: First submitted 2014-09-18; First posted 2014-09-22 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Organ Dysfunction Syndrome
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- APD probe (Experimental): Placement of a duodenal probe during 24 hours.
  Interventions: Device: APD probe

INTERVENTIONS:
Device: APD probe — The probe will be placed in the patient with an endoscopic procedure by a gastroenterologist (standard procedure for post-pyloric tubes placement).

SUMMARY:
For Intensive Care Units (ICU) patients, Multiple Organ Dysfunction Syndrome (MODS) is a very common complication yielding high morbidity and mortality. Inadequate regional perfusion of certain organs (gut, kidney, liver, etc) often caused by shock is the main cause of MODS. Current practice uses cardiac output data and blood pressure to manage shock but there are still lacks of information about the regional perfusion. This leads to late MODS diagnostics preventing the implementation of adequate treatment.

Gut perfusion monitoring seems to be a good target to assess the microcirculation but, nowadays, no practical methods or devices are available to measure the gut perfusion, and the current monitoring methods are not specific (CO, BP, OPS-SDF, PCO2, etc).

"MC Monitor" trial is a prospective, multi-center pilot study, enrolling 10 patients.

The probe will be used by intensivists on ICU patients with a risk of shock and requiring mechanical ventilation.

The probe will be placed in the patient with an endoscopic procedure by a gastroenterologist (standard procedure for post-pyloric tubes placement). This procedure will be used to assess the status of the gut mucosa prior to the placement of the APD probe.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or more,
* Male or female,
* ICU patient, on vasoactive amines, under mechanical ventilation,
* Stable hemodynamic status,
* Life expectancy expected to exceed 72 hours,
* Length of ICU stay greater than 5 days,
* Willing to participate and signed informed consent,
* Affiliation to the French social security system.

Exclusion Criteria:

* Pregnant or lactating woman,
* Ongoing enteral nutrition,
* Risk of gastrointestinal ischemia,
* History of pharyngeal surgery surgery, esophageal surgery, radiotherapy of mediastinal area,
* Known ear-nose-throat malignant disease,
* Unexplored dysphagia,
* Known recent gastrointestinal suture,
* Esophageal varices,
* Abdominal pain,
* Unstable cervical fracture,
* Moribund patient,
* Active participation in another investigational protocol within the past 30 days,
* Subject legally protected, under legal guardianship, deprived of his/her liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Absence of duodenal lesions | 24 hours
  Duodenal lesions are defined as visible alterations of the duodenum.

SECONDARY OUTCOMES:
Signal-to-noise ratio of the APD probe | 24 hours
  The signal is a reflect of the pulsatile flow in the duodenum. This assertion is evaluated thanks to a signal-to-noise ratio of the cardiac frequency in the PPG on other non-filtered signal componants.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Allaouchiche, Prof., Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - CHU Estaing - Service réanimation adultes, Clermont-Ferrand
  - Centre Hospitalier Lyon-Sud, Lyon
  - GHU Caremeau - Unité REA, Nîmes